CLINICAL TRIAL: NCT01675622
Title: A Comparative Study of Immediate-Release Oxycodone Capsules Versus Immediate-Release Morphine Tablets for the Treatment of Chinese Patients With Cancer Pain.
Brief Title: Immediate-Release Oxycodone Capsules Study in Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXYC10-CN-303
Record Dates: First submitted 2012-04-25; First posted 2012-08-30 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Cancer
Keywords: Cancer Pain
MeSH Terms: conditions — Neoplasms; Cancer Pain | interventions — Oxycodone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxycodone Capsules for cancer pain (Experimental)
  Interventions: Drug: Oxycodone
- Morphine tablets for cancer pain (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Oxycodone — dosage: 5mg, l0mg and 20mg dosage form: capsule frequency: every 6h, duration: 5-8 days
  Other Names: No other name in this study
  Arms: Oxycodone Capsules for cancer pain
Drug: Morphine — Morphine tablets 10mg and 20mg, oral every 4-6 hours
  Other Names: No other name
  Arms: Morphine tablets for cancer pain

SUMMARY:
The efficacy of dose titration of OxyNorm™(Oxycodone) immediate-release capsules versus morphine immediate-release tablets in the treatment of cancer pain.

DETAILED DESCRIPTION:
To compare the efficacy of dose titration of OxyNorm™(Oxycodone) immediate-release capsules versus morphine immediate-release tablets in the treatment of cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged 18 to 80 years inclusive, who with cancers of all type.
2. Patients with moderate to severe cancer pain, whose pain intensity Numeric Rating Scale ≥4.
3. Patients who can understand and are able to complete Numeric Rating Scale and Brief Pain Inventory assessment.
4. Patients who have given written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who are pregnant, or lactating.
2. Patients who are unable to manage their pain effectively with opioids.
3. Patient who need ≥120mg morphine or equivalent for treatment of pain at time of study entry;
4. Patients who are receiving chemotherapy, or still under the responsive period of chemotherapy (patients who are at the interval period of chemotherapy can be enrolled into study. That is to say, patients who completed chemotherapy for more than 2 weeks can enrolled, or patients has completed chemotherapy for at least one week could be enrolled at the discretion of the investigator).
5. Patients who have received radio-therapy for bony metastasis, patients receiving radiotherapy within the 4 week period before study entry (patient receiving radiotherapy for area other than pain area can be enrolled) , or patients who were scheduled to receive radiotherapy for pain area during study period.
6. Patients are receiving or should receive anti-convulsion drugs/anti- depression drugs considered by investigator for the treatment of neuropathy pain. Patients are receiving or should receive any analgesic other than study medicine, which including NSAIDs.
7. Patients with other unstable disease, or with dysfunction of important organ.
8. Patients with an ongoing infection, abscess or fever.
9. Patient with serious abnormal liver/ renal function (ALT/Aspartate Transaminase/creatinine/urea nitrogen) which is higher than 3 times of upper limit;
10. Paralytic or mechanical ileus;
11. Persistent asthma, chronic obstructive diseases, and cor pulmonary;
12. Intracranial neoplasms, and intracranial hypertension with central respiratory depression risk.
13. Monoamine oxidase inhibitors (MAOIs) or same type drugs have been administered in last 2 weeks;
14. Patients who are currently taking active treatment for epilepsy or arrhythmias.
15. Patients with known sensitivity or record of specific or allergic reaction to oxycodone or morphine.
16. Patients excluded by the contra-indications, adverse drug reaction (ADRs) and drug interactions of oxycodone or morphine as detailed in the data sheet, summary of product characteristics or investigator's brochure.
17. Patients with a history of drug or alcohol abuse.
18. Patients who participated in another clinical research study involving a new chemical entity within one month prior to study entry.
19. Patients whose concomitant medication is likely to be changed within the study period, with the exception of treatment for opioid side effects.
20. Patients who, in the opinion of the investigator, are unsuitable to participate in the study for any other reason not mentioned in the inclusion and exclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shiying Yu, Prof., Principal Investigator — Wuhan TongJi Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 242 subjects were enrolled from 20 centers in which 192 subjects completed the study and 50 subjects did not completed the study. All the subjects were recruited from medical clinic.The recruitment period is from 2011 Jan to 2012 Mar.
Pre-assignment Details: Patients with moderate to severe cancer pain requiring oral opioid therapy were screened. All the patients who meets the inclusion/exclusion criteria were enrolled to double blind treatment phase. No wash our or run-in period required by protocol.
Groups:
- Oxycodone Capsules for Cancer Pain: Oxycodone: dosage: 5mg, l0mg and 20mg dosage form: capsule frequency: every 6h, duration: 5-8 days. All patients completed the double-blind treatment entered into period 2.
  period 2 is open treatment phase. Patients received two weeks treatment of oxycodone hydrochloride controlled-release tablets.
- Morphine Tablets for Cancer Pain: Morphine: Morphine tablets 10mg and 20mg, oral every 4-6 hours. All patients completed the double-blind treatment entered into period 2.
  period 2 is open treatment phase. Patients received two weeks treatment of oxycodone hydrochloride controlled-release tablets.
Period: Overall Study
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Started | 122 | 120
Completed | 96 | 96
Not Completed | 26 | 24
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 12 | 10
Not completed — Protocol Violation | 4 | 1
Not completed — Lack of Efficacy | 2 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Other | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain | Total
Number analyzed (Participants) | 120 | 118 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.62 (12.96) | 57.05 (12.07) | 56.83 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 62 | 59 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 119 | 117 | 236
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 120 | 118 | 238
height [Mean (Standard Deviation); unit: centimeter] | 164.5 (7.45) | 164.99 (8.20) | 164.74 (7.82)
weight [Mean (Standard Deviation); unit: kg] | 58.64 (10.79) | 58.34 (11.01) | 58.49 (10.88)

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS)
Description: The numerical rating scale is the tool to assess pain level using a numerical rating scale. The primary outcome measurement is the average change of NRS score after double blind treatment between the two treatment groups. The NRS evaluates the pain level using number scale from 0 to 10. 0 means not painful and 10 means extremely painful. 1 to 3 is lightly pain, 4-6 is moderate pain and 7 to 10 is severe pain. There is no subscales used for NRS reporting.
Time Frame: baseline up to 5-8 days (double blind period)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
scores on a scale | 3.91 (2.31) | 3.87 (2.22)

2. Secondary Outcome: The Average Dose of Study Medicine Used During Double Blind Treatment Period
Description: the average dose of study medicine used during double blind treatment period between the two treatment groups.
Time Frame: baseline up to 5-8 days (double blind period)
Population: The average total dosage during double-blind treatment was defined as a primary efficacy endpoint in the protocol, but this study was a non-inferiority study, and non-inferiority analysis could not be performed in average total dosage in data processing and statistics.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
mg
  Average total dosage during double-blind titration | 83.29 (82.87) | 141.61 (112.10)
  Ave. total dosage during double-blind maintenance | 167.41 (103.92) | 308.63 (189.93)

3. Secondary Outcome: Brief Pain Inventory (BPI) Change From Baseline to After Double Blind Period
Description: The secondary outcome measurement is the change between BPI score at baseline and after completion of double blind treatment between the two treatment groups. The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning. This tool measures the worst/least pain in the passed 24 hours, and the average/current pain in last 24 hours. The scale is numerically from 0 to 10. 0 means not painful, 10 means extremely painful. The BPI is the average number of above 4 BPI Pain Items.
Time Frame: baseline up to 5-8 days (double blind period)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
scores on a scale
  Highest pain intensity in 24 hrs | 4.25 (1.98) | 4.03 (2.20)
  Lowest pain intensity in 24 hrs | 2.62 (2.08) | 2.53 (1.98)
  Average pain intensity in 24 hrs | 3.39 (1.80) | 3.35 (1.73)
  Current Pain intensity | 3.78 (1.94) | 3.70 (1.88)

4. Secondary Outcome: Times of Breakthrough Pain Occurrence
Description: the times of breakthrough pain occurrence during double blind treatment phase between the two treatment groups
Time Frame: Within 8 days after baseline
Measure: Number; unit: breakthrough pain events
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
breakthrough pain events | 15 | 20

5. Secondary Outcome: Patient Assessments of Satisfaction for Pain Management
Description: the number of patients of satisfaction for pain management between the two treatment groups at the end of double blind treatment and the open label treatment period.
Time Frame: baseline up to 19-22 days (open label treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
Participants
  Very satisfied | 35 | 37
  Satisfied | 64 | 61
  Neutral | 9 | 5
  Dissatisfied | 1 | 4
  Missing | 11 | 11

6. Secondary Outcome: Average Number of Titrations
Description: the average times to change the dose in order to find the proper dose between two treatment groups
Time Frame: baseline up to 1-3 days(double blind period)
Population: Dosing change frequency for complete titration
Measure: Mean (Standard Deviation); unit: dose changes
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
dose changes | 8.25 (4.52) | 7.89 (3.43)

7. Secondary Outcome: Brief Pain Inventory (BPI) Change From Baseline to Open Label Treatment
Description: The secondary outcome measurement is the change of BPI score from baseline to the end of open label treatment between the two treatment groups. The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning. This tool measures the worst/least pain in passed 24 hours, and the average/current pain in last 24 hours. The scale is numerically from 0 to 10. 0 means not painful, 10 means extremely painful. The BPI is the average number of above 4 BPI Pain Items.
Time Frame: baseline up to 19-22 days (open label treatment)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
scores on a scale
  Highest pain intensity in 24 hrs | 3.98 (2.09) | 3.95 (1.92)
  Lowest pain intensity in 24 hrs | 2.57 (2.05) | 2.64 (1.98)
  Average pain intensity in 24 hrs | 3.33 (1.83) | 3.48 (1.57)
  Current Pain intensity | 3.62 (1.87) | 3.71 (1.57)

8. Secondary Outcome: the Total Dose of Rescue Medicine for Breakthrough Pain.
Description: the total dose of rescue medicine for breakthrough pain during double blind phase between the two treatment groups
Time Frame: baseline up to 22 days (double blind period)
Population: The double-blind titration period was the dose adjusting phase, so breakthrough pain occurrences in this period were not included in statistical analysis. After titration was completed, subjects entered into maintenance treatment with the titrated dose.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
mg
  the total dose of rescue medicine -day1 | 10.63 (7.76) | 7.00 (4.83)
  the total dose of rescue medicine -day2 | 10.00 (8.29) | 6.00 (2.07)
  the total dose of rescue medicine-day3 | 10.63 (8.21) | 6.82 (2.52)
  the total dose of rescue medicine-day4 | 20.00 (8.94) | 7.86 (3.93)
  the total dose of rescue medicine-day5 | 11.00 (10.84) | 6.67 (4.08)
  the total dose of rescue medicine -day6 | 0 (0) | 5.00 (0.00)
  the total dose of rescue medicine after day6 | 5.00 (0) | 5.00 (0.00)

9. Secondary Outcome: Degree of Pain Relief Within 24hrs After Treatment
Description: Brief Pain Inventory (BPI) Change From Baseline to After Double Blind Period. The BPI is the average number of above 4 BPI Pain Items. For the degree of pain relief within 24hrs after treatment, 0 means zero relief and 100 means completely relief with unit of percentage(%).
Time Frame: baseline up to 5-8 days (double blind period)
Measure: Mean (Standard Deviation); unit: percentage of pain relief
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
percentage of pain relief | 35.23 (28.27) | 34.19 (30.85)

10. Secondary Outcome: Brief Pain Inventory (BPI) Change From Baseline to Open Label Treatment
Description: For the degree of pain relief within 24hrs after treatment, 0 means zero relief and 100 means completely relief with unit of percentage(%).
Time Frame: baseline up to 19-22 days (open label treatment)
Measure: Mean (Standard Deviation); unit: percentage of pain relief
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
Number analyzed (Participants) | 120 | 118
percentage of pain relief | 32.31 (30.80) | 31.64 (29.73)

ADVERSE EVENTS:
Time Frame: up to 36 days
Description: The AE collection period including maximally 7 days screening and 5 to 8 days double blind period, and then 14 days open treatment period. 7 days safety follow up.
Arm/Group | Oxycodone Capsules for Cancer Pain | Morphine Tablets for Cancer Pain
All-Cause Mortality (participants affected / at risk) | 2/120 | 2/118
Serious Adverse Events (participants affected / at risk) | 4/120 | 2/118
Other Adverse Events (participants affected / at risk) | 76/120 | 75/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone Capsules for Cancer Pain (N=120) | Morphine Tablets for Cancer Pain (N=118)
Respiratory and circulatory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — 4 patients died of respiratory/circulatory failure due to progression of the underlying disease, which were not related to the study drug determined by the investigator
ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) — 1 patient had ileus, which was possibly related to the study drug determined by the investigator, and the associated symptoms completely disappeared at the end of follow-up period.
Brain metastases (Nervous system disorders) | 1 (1) | 0 (0) — 1 patient was hospitalized for brain metastases, which was unrelated to the study drug determined by the investigator, and the associated symptoms still persisted at the end of follow-up period;
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone Capsules for Cancer Pain (N=120) | Morphine Tablets for Cancer Pain (N=118)
Constipation (Gastrointestinal disorders) | 38 (41) | 43 (47)
Nausea (Gastrointestinal disorders) | 25 (31) | 26 (30)
Vomiting (Gastrointestinal disorders) | 25 (27) | 24 (25)
Dizziness (Nervous system disorders) | 9 (10) | 6 (6)
Fever (Immune system disorders) | 8 (9) | 4 (6)
Drowsiness (Nervous system disorders) | 8 (8) | 4 (4)
Loss of appetite (Nervous system disorders) | 5 (5) | 3 (3)
Fatigue (Psychiatric disorders) | 4 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Low platelet count (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No